CLINICAL TRIAL: NCT02761109
Title: Postoperative Renal, Pulmonary, Cardiovascular Complications and Use of Blood Components in Patients Undergoing Liver Transplantation
Brief Title: Postoperative Complications After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Giorgio Della Rocca, Full Professor, Azienda Ospedaliera S. Maria della Misericordia
Other Study IDs: OLTXCompl
Record Dates: First submitted 2016-04-21; First posted 2016-05-04 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Liver Transplantation; Postoperative Renal Complication; Postoperative Pulmonary Complication; Postoperative Cardiovascular Complication; Blood Components Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Incidence and risk factors for renal, cardiovascular and pulmonary complications after liver transplantation are not well defined. Blood products requirement is an important aspect of orthotropic liver transplantation (OLTx) management and has a great impact on patient's outcome. Transfusions of blood products increase perioperative complications and reduce graft and patients survival.

The primary endpoint of the study is to evaluate the incidence of renal complication during ICU stay after liver transplantation using RIFLE criteria; secondary endpoint is to evaluate the incidence of cardiovascular and pulmonary complications. In addition patients' survival and the relationship between blood components use with the development of post-operative complications are evaluated.

DETAILED DESCRIPTION:
It is conducted a prospective observational cohort study in all Italian liver transplant centers. Adult (> 18 years old) recipients of deceased liver graft between January 2011 and December 2013 were eligible for inclusion. Exclusion criteria were the use of living organ donation, retransplantation, pediatric transplantations, combined transplantation and fulminant hepatic failure.

Investigators collected data using a prospectively maintained computer database managed by the Italian Ministry of Health "Centro Nazionale Trapianti". Anesthetic and perioperative management followed the routine local institution protocols.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more

Exclusion Criteria:

* Age less than 18 years;
* Liver transplantation living related donor;
* Retransplantation;
* combined transplantation;
* fulminant hepatic failure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years old or more undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Incidence of renal complication after liver transplantation | At 72 post operative hours
  The primary endpoint of the study is to evaluate the incidence of renal complication during ICU stay after liver transplantation using RIFLE criteria

SECONDARY OUTCOMES:
Incidence of cardiovascular complication after liver transplantation | During ICU length of stay, an average of 4 days.
  To evaluate the incidence of postoperative cardiovascular complications
Incidence of pulmonary complication after liver transplantation | During ICU length of stay, an average of 4 days.
  To evaluate the incidence of postoperative pulmonary complications
Number of patients alive after liver transplantation that required blood components transfusion | At 1 year and at 3 years after liver transplantation
  To investigate the relationship of cardiovascular, pulmonary, renal complications after liver transplantation and the blood components consumption with mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica di Anestesia, rianimazione e terapia intensiva, Udine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Watt KD, Pedersen RA, Kremers WK, Heimbach JK, Charlton MR. Evolution of causes and risk factors for mortality post-liver transplant: results of the NIDDK long-term follow-up study. Am J Transplant. 2010 Jun;10(6):1420-7. doi: 10.1111/j.1600-6143.2010.03126.x. Epub 2010 May 10. PMID 20486907
- [Result] Barri YM, Sanchez EQ, Jennings LW, Melton LB, Hays S, Levy MF, Klintmalm GB. Acute kidney injury following liver transplantation: definition and outcome. Liver Transpl. 2009 May;15(5):475-83. doi: 10.1002/lt.21682. PMID 19399734
- [Result] Fouad TR, Abdel-Razek WM, Burak KW, Bain VG, Lee SS. Prediction of cardiac complications after liver transplantation. Transplantation. 2009 Mar 15;87(5):763-70. doi: 10.1097/TP.0b013e318198d734. PMID 19295324
- [Result] Levesque E, Hoti E, Azoulay D, Honore I, Guignard B, Vibert E, Ichai P, Antoun F, Saliba F, Samuel D. Pulmonary complications after elective liver transplantation-incidence, risk factors, and outcome. Transplantation. 2012 Sep 15;94(5):532-8. doi: 10.1097/TP.0b013e31825c1d41. PMID 22885879
- [Result] Ramos E, Dalmau A, Sabate A, Lama C, Llado L, Figueras J, Jaurrieta E. Intraoperative red blood cell transfusion in liver transplantation: influence on patient outcome, prediction of requirements, and measures to reduce them. Liver Transpl. 2003 Dec;9(12):1320-7. doi: 10.1016/jlts.2003.50204. PMID 14625833